CLINICAL TRIAL: NCT06652906
Title: A Prospective, Multicenter, Randomized Controlled Clinical Trial on the Safety and Efficacy of Sodium Phosphate Powder for Intestinal Preparation in the Population Aged 50 to 70 Years Old
Brief Title: Study on the Safety and Efficacy of Sodium Phosphate Powder for Intestinal Preparation in People Aged 50 to 70 Years Old
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: LY-2024-062-B
Record Dates: First submitted 2024-06-11; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Physical Examination

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sodium phosphate powder group (Experimental): Sodium phosphate powder group: After admission, patients will undergo comprehensive renal function and electrolyte tests. The first medication will be taken at 7pm the day before the examination. One bag of sodium phosphate powder will be diluted with 800ml or more of warm and cool water before taking. The second dose of medication should be taken at 7am on the day of operation or examination (or at least 3 hours before the examination), with the same usage as the first dose, with a 12 hour interval between each dose. The standard dose for each dose is 1 bag, until clear water like stool appears.
  Interventions: Drug: Sodium phosphate powder
- Polyethylene glycol electrolyte dispersion (Active Comparator): Polyethylene glycol electrolyte powder group: After admission, the patient underwent comprehensive renal function and electrolyte examination. The evening before the intestinal examination, 2000ml of polyethylene glycol electrolyte powder III isotonic solution was taken, 250ml every 10-15 minutes, and it was taken within 2 hours. On the day of examination, 2000ml of polyethylene glycol electrolyte powder III isotonic solution was taken again 3-4 hours in advance until clear water like stool appeared.
  Interventions: Drug: Polyethylene glycol electrolyte dispersion

INTERVENTIONS:
Drug: Sodium phosphate powder — After admission, the patient underwent comprehensive renal function and electrolyte tests. The first medication was taken at 7pm the day before the examination. One bag of sodium phosphate powder was diluted with 800ml or more of warm and cool water before taking. The second dose of medication should be taken at 7am on the day of operation or examination (or at least 3 hours before the examination), with the same usage as the first dose, with a 12 hour interval between each dose. The standard dose for each dose is 1 bag, until clear water like stool appears.
  Arms: Sodium phosphate powder group
Drug: Polyethylene glycol electrolyte dispersion — After admission, the patient underwent comprehensive renal function and electrolyte examination. The evening before the intestinal examination, 2000ml of polyethylene glycol electrolyte San III isotonic solution was taken, 250ml every 10-15 minutes, and it was taken within 2 hours. On the day of examination, 2000ml of polyethylene glycol electrolyte San III isotonic solution was taken 3-4 hours in advance until clear water like stool appeared.
  Other Names: Fortrans
  Arms: Polyethylene glycol electrolyte dispersion

SUMMARY:
Project Name: Safety and Efficacy of Sodium Phosphate Powder for Intestinal Preparation in People Aged 50 to 70: A Prospective, Multicenter, Randomized Controlled Clinical Trial The main purpose of the study is to investigate the effectiveness and safety of sodium phosphate powder for intestinal preparation in people aged 50 to 70.

Secondary objective: To study the tolerance of sodium phosphate powder for intestinal preparation in the population aged 50 to 70 years and its impact on The impact of lesion detection. A prospective multicenter intervention randomized controlled clinical study of research design The total number of cases is 362 in the group leader center, with a total of 8 participating centers each having 44 cases.

Treatment plan: Sodium phosphate powder group or Fujingqing group

Main efficacy evaluation indicators:

The effective rate of intestinal preparation, that is, the endoscopist determines that the patient's Boston intestinal preparation score is ≥ 6 points and The ratio of patients with a bowel preparation score of ≥ 2 points per segment to the total number of patients.

Safety evaluation indicators Adverse reaction incidence rate Statistical methods: Numerical variables are described using mean ± standard deviation (Mean ± SD) and estimated using normal distribution method

Analysis of main efficacy indicators:

Based on the intention to treat set, including all qualified patients undergoing colonoscopy, efficacy evaluation will be conducted, Use chi square test or Fisher's exact probability method for inter group comparison. The inspection level is 0.05.

Research period from April 2023 to August 2024

DETAILED DESCRIPTION:
Project Name: Safety and Efficacy of Sodium Phosphate Powder for Intestinal Preparation in People Aged 50 to 70: A Study Prospective, multicenter, randomized controlled clinical trials The main purpose of the study is to investigate the effectiveness and safety of sodium phosphate powder for intestinal preparation in people aged 50 to 70 years old Completeness. Secondary objective: To study the tolerance of sodium phosphate powder for intestinal preparation in the population aged 50 to 70 years and its impact on The impact of lesion detection. A prospective multicenter intervention randomized controlled clinical study of research design The total number of cases is 362 in the group leader center, with a total of 8 participating centers each having 44 cases.

Case selection Inclusion Criteria

1. Age range from 50 to 70 years old, regardless of gender;
2. No contraindications for colonoscopy examination, plan to undergo colonoscopy examination in the near future;
3. Agree to participate in this study. Exclusion criteria

1. Patients with a history of colorectal surgery (resection of malignant tumors, resection of colorectal perforation, etc.); 2. Electrolyte disorders and hemodialysis patients; 3. Patients with active lower gastrointestinal bleeding; 4. Patients with abnormal coagulation function; 5. Concomitant severe primary diseases such as lung, liver, kidney, and hematopoietic system, liver function ALT AST Exceeding the upper limit of the reference value by 1.5 times, or Cr exceeding the upper limit of the reference value; 6. Merge other diseases that may affect the efficacy judgment or pose a significant risk, such as inflammatory bowel disease Acute phase, colon cancer, intussusception, volvulus, intestinal obstruction, peritonitis, ascites, refractory Constipation, etc; 7. Patients with mental illness and severe neurosis; 8. Patients who are known to have allergies to the investigational or control drugs; 9. Those who have participated in other clinical studies within one month; 10. Researchers believe that there are other situations that are not suitable for inclusion, and patients are unwilling to be included in the study.

Version number: 3.0 Date: December 5th, 2023 two Treatment plan: Sodium phosphate powder group: Patients will receive comprehensive renal function and electrolyte tests after admission, and will take medication for the first time At 7pm the day before the inspection, 1 bag of sodium phosphate powder should be diluted with 800ml or more of warm and cool boiled water Take after release. The second medication should be taken at 7am on the day of operation or examination (or before the examination) Less than 3 hours), the usage is the same as the first time, with a 12 hour interval between each session. The standard dose for each session is 1 bag, Until clear water like stool appears, the patient should take a photo of their intestines to prepare for feces, and record the results of each dose taken The time of the first and last bowel movements, as well as the frequency of each bowel movement. After the intestinal preparation is completed, Further improvement of renal function and electrolyte examination, followed by colonoscopy examination and retention of operation video, necessary Take live tissue for examination when necessary. Fujingqing group: After admission, patients were given comprehensive renal function and electrolyte tests, and the day before intestinal examination Take 2000ml of polyethylene glycol electrolyte powder III isotonic solution at night, every 10-15 minutes 250ml, taken within 2 hours, take polyethylene glycol electrolyte powder III 3-4 hours in advance on the day of examination 2000ml of isotonic solution until clear water like stool appears, and the patient should take a photo of the intestine to prepare the stool, Record the time of the first and last bowel movements, as well as the frequency of bowel movements, after each dose of medication.

After completing the intestinal preparation, the renal function and electrolyte examination should be further improved, followed by a colonoscopy examination Retain operation videos and, if necessary, take live tissue for inspection. Efficacy evaluation Effectiveness evaluation indicators (primary and secondary efficacy indicators)

Main efficacy evaluation indicators:

The effective rate of intestinal preparation, that is, the endoscopist determines that the patient's Boston intestinal preparation score is ≥ 6 points and The ratio of patients with a bowel preparation score of ≥ 2 points per segment to the total number of patients.

Secondary efficacy evaluation indicators:

The effective rate of segmented intestinal preparation, i.e., according to the Boston score for the 3 segments of the colon (rectum sigmoid) Colon, transverse colon descending colon, ascending colon cecum) were scored separately.

Polyp detection rate, which is the ratio of patients with polyps detected by colonoscopy to the total number of patients.

Adenoma detection rate refers to the ratio of patients with adenomas detected by colonoscopy to the total number of patients.

Patient subjective tolerance score: including taste score and willingness to repeat use score.

Safety evaluation indicators The incidence of adverse reactions, namely nausea, vomiting, abdominal pain, and The proportion of patients with adverse reactions such as bloating and electrolyte imbalance to the total number of patients.

Statistical methods: Numerical variables are described using mean ± standard deviation (Mean ± SD) and estimated using normal distribution method Version number: 3.0 Date: December 5th, 2023 three Calculate the 95% bilateral confidence interval of the overall mean and use t-test for inter group comparison; Categorical variable Describe using frequency (n) and composition ratio (%), i.e. [n (%)], and estimate each using normal approximation method 95% confidence interval for the overall group rate, using chi square test or Fisher's exact probability method Compare between groups.

Analysis of main efficacy indicators:

Based on the intention to treat set, including all qualified patients undergoing colonoscopy, efficacy evaluation will be conducted, Use chi square test or Fisher's exact probability method for inter group comparison. The inspection level is 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Age 50 to 70 years old, gender unlimited
2. No contraindications for colonoscopy examination, planned to undergo colonoscopy examination in the near future
3. Agree to participate in this study

Exclusion Criteria:

1. Patients with a history of colorectal surgery (resection of malignant tumors, resection of rectal perforation, etc.)
2. Electrolyte disorders and hemodialysis patients
3. Patients with active lower gastrointestinal bleeding
4. Patients with abnormal coagulation function
5. Concomitant severe primary diseases such as lung, liver, kidney, and hematopoietic system, liver function ALT AST exceeds the upper limit of the reference value by 1.5 times, or Cr exceeds the upper limit of the reference value
6. Merge other diseases that may affect the efficacy judgment or pose a significant risk, such as acute inflammatory bowel disease, colon cancer, intussusception, volvulus, intestinal obstruction, peritonitis, ascites, stubborn constipation, etc
7. Patients with mental illness and severe neurosis
8. Patients known to have allergies to the investigational or control drugs
9. Participated in other clinical researchers within one month
10. Researchers believe that there are other situations that are not suitable for inclusion, and patients are unwilling to be included in the study

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2024-06-11 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Qualified rate of intestinal preparation | Within three months
  According to the Boston intestinal score, the evaluation was completed by a colonoscopy doctor.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Jiaotong University School of Medicine, Renji Hospital, Shanghai, Shanghai Municipality, China